CLINICAL TRIAL: NCT01564030
Title: Qualitative Ultrasound Assessment of the Gastric Content of Pregnant Women at Term
Brief Title: Gastric Ultrasound in Pregnant Women at Term
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 12-01
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Respiratory Aspiration; Pregnancy
Keywords: Pregnancy; Respiratory aspiration; Gastric contents; Ultrasound
MeSH Terms: conditions — Respiratory Aspiration | interventions — Fluid Therapy; Polymethyl Methacrylate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Empty stomach (Other): Patients have fasted for 8 hours.
  Interventions: Other: Empty
- Fluid (Other): Patients have fasted for 8 hours, followed by the consumption of 250mL of apple juice.
  Interventions: Other: Fluid
- Solid (Other): Patients have fasted for 8 hours, followed by the consumption of their breakfast.
  Interventions: Other: Solid

INTERVENTIONS:
Other: Empty — overnight fast
  Arms: Empty stomach
Other: Fluid — 250mL apple juice
  Arms: Fluid
Other: Solid — breakfast
  Arms: Solid

SUMMARY:
Solid food or fluid residue in the stomach is always a major concern when patients need medical procedures under sedation or general anesthesia, due to the high risk of pulmonary aspiration of the stomach contents. This is especially important in emergency procedures, when a fasting period is not observed. The aspiration of the stomach contents into one's lungs can lead to serious complications (such as severe respiratory failure). Information from a bedside ultrasound assessment of the stomach may be a very useful tool to decide whether or not it's safe to proceed, cancel or delay a surgical procedure.

DETAILED DESCRIPTION:
Food residue in the stomach of patients scheduled to have surgery is considered a major risk factor for pulmonary aspiration of gastric contents. The resulting respiratory compromise after aspiration is associated with significant morbidity and mortality. The risk of pulmonary aspiration is especially important in pregnant women, as they may often require surgery without having observed appropriate fasting. A bedside ultrasound assessment fo the status of the gastric content would be of great value for the clinician. This technique has recently been shown very promising in non-pregnant patients and it is important to study its feasibility in the pregnant population.

In this study, patients fast overnight and are randomized to the following groups: empty, fluid (250 mL of apple juice before scanning) or solid (full breakfast). Their gastric contents are then assessed by 3 different anesthesiologists, using ultrasound. At the end of the scanning, the true stomach contents are revealed. The ability of the assessors to accurately predict stomach contents, as well as the inter-observer agreement, will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer non-laboring pregnant women >32 weeks gestation
* 18 years or older
* ASA status I-III
* Weigh between 50 and 120kg
* Height at least 150cm or taller
* Written informed consent

Exclusion Criteria:

* Known pre-existing abnormal anatomy of the upper GI tract
* Protocol violation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Reliability of the ultrasonographic diagnosis of the gastric status | 30 minutes
  Three physicians trained in gastric ultrasound will be blinded to the treatment group the patient was in, perform an ultrasound, and try to guess whether the patient has an empty stomach, consumed fluids only, or consumed a full meal.

SECONDARY OUTCOMES:
Inter-observer agreement of gastric content diagnosis | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Arzola C, Cubillos J, Perlas A, Downey K, Carvalho JC. Interrater reliability of qualitative ultrasound assessment of gastric content in the third trimester of pregnancy. Br J Anaesth. 2014 Dec;113(6):1018-23. doi: 10.1093/bja/aeu257. Epub 2014 Jul 30. PMID 25080428